CLINICAL TRIAL: NCT03995797
Title: Randomised, Sham Controlled Trial of Fotona Smooth Erbium Yag Laser In the Treatment of Pelvic Organ Prolapse.
Brief Title: VESPER: Pelvic Organ Prolapse Study
Acronym: VESPER:POP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not open
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-FAM-02
Record Dates: First submitted 2019-03-28; First posted 2019-06-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Active Comparator): Treatment with erbium YAG laser
  Interventions: Procedure: Laser therapy
- Sham arm (Placebo Comparator): Sub therapeutic procedure with erbium YAG laser
  Interventions: Procedure: Laser therapy

INTERVENTIONS:
Procedure: Laser therapy — Erbium YAG laser

SUMMARY:
Patients seen with Stage 1-2 pelvic organ prolapse (POP) who have failed conservative treatments will be offered to participate in a sham controlled RCT of outpatient therapy with the Fotona Smooth Erbium Yag Laser. Patients will be randomised to either outpatient laser treatments or sham treatments. Patients will be blinded to which arm they have been randomised. Patients will be asked to complete appropriate relevant symptom and quality of life questionnaires and prolapse scoring, prior to treatment and at each monthly treatment and then 6 and 12 months following the final treatment. At 6 months following final treatment, Sham patients will be un-blinded and offered the laser therapy if they wish.

DETAILED DESCRIPTION:
All patients with symptomatic stage 1-2 POP, who have failed / declined conservative therapy will be informed about the study and invited to participate.

Once eligibility for inclusion into the study has been confirmed and written consent has been obtained, the patient will be invited for a baseline visit. At this visit the patient will have their medical history confirmed and have all Pelvic Organ Prolapse Quantification Score (PoP-Q) measurements made. They will be given the ICIQ Vaginal Symptom (ICIQ-VS) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) questionnaire.

Patients will be randomised and blinded to their allocated arm: active treatment or sham treatment (2:1, treatment : Sham).

Patients will then undergo 4 outpatient treatment visits. The timing of visits will be from 1 month apart. Before each treatment, they will have their urine tested for infection (dipstick urinalysis) and a pregnancy test (not required if had hysterectomy / sterilised). If urinalysis is negative, they will be receive an outpatient ProlapLase treatment which lasts 20 minutes. They will be given a leaflet outlining what to expect and a contact number if they have any concerns or questions. They will be asked about any deleterious effects since their last appointment, have a PoPQ score recorded and asked to complete a Patient Global Impression of Improvement (PGI-I) questionnaire. Patients will routinely receive 4 treatments. Each treatment will be 4 weeks apart.

Patients will be invited to attend a follow up visit 6 months after the 4th treatment. They will be asked if they are happy to continue to participate in the trial and if happy, asked to complete International Consultation on Incontinence Questionnaire (ICIQ-VS), Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) and Patient Global Impression of Improvement (PGI-I) symptom questionnaires and undergo a Pelvic Organ Prolapse Quantification Score (PoP-Q) score. Patients will be asked about any Adverse Event / Serious Adverse Event since involvement in the study. Patients randomised to the Sham arm will be un-blinded at 6 months and offered the treatments (x4) if they wish. They will then be followed up at 6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria

1. Adult Female, 18 years of age or older
2. Clinical diagnosis of symptomatic stage 1-2 pelvic organ prolapse (PoPQ classification)
3. Failed / declined conservative treatments, such as pelvic floor muscle training or vaginal pessaries

Exclusion Criteria:

Exclusion Criteria

1. Pre-existing bladder pathology including prior radiation treatment
2. Pregnancy
3. BMI>35
4. Radical pelvic surgery or previous incontinence surgery
5. Urinary tract infection or other active infections of urinary tract or bladder
6. Any form of pelvic organ prolapse greater than stage 2, according to POP-Q
7. Diagnosis of collagen disorders eg.benign joint hypermobility / Elhers-Danlos / Marfans etc.
8. Incomplete bladder emptying
9. Vesicovaginal fistula
10. Faecal incontinence
11. Unwillingness or inability to complete follow-up schedule
12. Unwillingness or inability to give Informed Consent
13. Failure to comply with diary requirements during extended baseline period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification Score (POP-Q) between baseline and 6 months after treatment. | 6 months
  The change in Pelvic Organ Prolapse Quantification Score (PoP-Q)classification between baseline and 6 months, range = 0 - stage 4
Pelvic Organ Prolapse Quantification Score (POP-Q) between baseline and 12 months after treatment. | 12 months
  The change in Pelvic Organ Prolapse Quantification Score (PoP-Q) classification between baseline and 12 months, range = 0 - stage 4

SECONDARY OUTCOMES:
Change in mean International Consultation on Incontinence Questionnaire - Vaginal Symptoms (ICIQ-VS) test scores from baseline to 6 months post treatment | 6 months
  Change in mean test scores from baseline to 6 months post treatment. Range:
  vaginal symptom scores (0-53), sexual matters scores (0-58), quality of life scores (0-10); higher score indicates greater severity of symptoms.
Change in mean International Consultation on Incontinence Questionnaire - Vaginal Symptoms (ICIQ-VS) test scores from baseline to 12 months post treatment | 12 months
  Change in mean test scores from baseline to 12 months post treatment. Range:
  vaginal symptom scores (0-53), sexual matters scores (0-58), quality of life scores (0-10); higher score indicates greater severity of symptoms.
Patient's Global Impression of Improvement (PGI-I) at 6 months | 6 months
  Questionnaire scores - range 1 (very much worse) to 7 (very much improved)
Patient's Global Impression of Improvement (PGI-I) at 12 months | 12 months
  Questionnaire scores - range 1 (very much worse) to 7 (very much improved)
Change in mean Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) scores | 6 months
  Change in mean test scores - range = 0 - 48; Higher value = increased sexual function, lower value = less sexual function
Change in mean Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) scores | 12 months
  Change in mean test scores - range = 0 - 48; Higher value = increased sexual function, lower value = less sexual function
Pain visual analogue scale | 4 months
  Patient reported assessment of pain on 10cm visual analogue scale during treatment, range 1 - 10cm; 0= no pain, 10= severe pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601